CLINICAL TRIAL: NCT04423445
Title: Laser Acupuncture Combined With Acupressure Improves Low Back Pain and Quality of Life: a Randomized Controlled Trial
Brief Title: Laser Acupuncture and Acupressure for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, Hsueh-Hua Yang, Principal Investigator, En Chu Kong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECKIRB1071102
Record Dates: First submitted 2020-04-18; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Low Back Pain
Keywords: Acupuncture; acupressure; low back pain; low-level laser; life dysfunction; hospital nurses
MeSH Terms: conditions — Low Back Pain | interventions — Acupressure; Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: This single-blinded randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture combined with acupressure (LAA) (Experimental): A 4-week LAA intervention included low-level laser acupuncture and auricular acupressure. Six acupuncture points were selected, and three auricular points. Participants received laser acupuncture on the six selected acupuncture points bilaterally twice a week for 4 weeks. A seed was taped onto each of the three points of the unilateral ear (initially, the left ear), where it remained for five days. Pressing on each of the seeds for one minute three times a day was required, but the stimulation intensity was adjusted depending on the participant's individual tolerance. After five days, the seed was removed, and a new seed was taped on the other ear.
  Interventions: Other: Laser acupuncture combined with acupressure
- Control group (No Intervention): Control participants received a similar intervention, but without laser energy output or acupressure.

INTERVENTIONS:
Other: Laser acupuncture combined with acupressure — Participants received laser acupuncture on the six selected acupuncture points bilaterally twice a week for 4 weeks. A seed was taped onto each of the three points of the unilateral ear (initially, the left ear), where it remained for five days. Pressing on each of the seeds for one minute three times a day was required, but the stimulation intensity was adjusted depending on the participant's individual tolerance. The de qi sensation appears to be an established intervention efficacy indicator during auricular acupressure. After five days, the seed was removed, and a new seed was taped on the other ear.
  Other Names: Control group
  Arms: Laser acupuncture combined with acupressure (LAA)

SUMMARY:
Background: Low back pain (LBP) is a common, huge health and socioeconomic health problem that affects physiological functions and reduces work efficiency in nurses.

Objective: This study aimed to evaluate the effect of low-level laser acupuncture combined with acupressure (LAA) on pain intensity, pain interference and life dysfunction in hospital nurses with LBP.

Methods: This single-blinded randomized controlled trial enrolled a convenience sample of nurses from one teaching hospital. Seventy-six participants were randomly assigned to the LAA group (n=38) receiving low-level laser acupuncture and auricular acupressure for four weeks, and a control group (n=38) receiving a similar intervention but without laser energy and acupressure. Data were collected using the Short Form of the Brief Pain Inventory (BPI-SF) and Roland-Morris Disability Questionnaire (RDQ) at three time points: baseline before the intervention, and Week 2 and Week 4 during the intervention.

DETAILED DESCRIPTION:
The enrollment criteria were age more than 20 years, low back pain with visual analogue scale (LBP_VAS) ≧3, no regular treatment for low back pain within six weeks, and willing to participate in this study. Exclusion criteria were open wounds on lower back, tumor on the back, ankylosing spondylitis, previous lumbar surgery, coagulopathy or bleeding tendency, or pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* age more than 20 years, low back pain with visual analogue scale (LBP_VAS) ≧3
* no regular treatment for low back pain within six weeks
* willing to participate in this study

Exclusion Criteria:

* open wounds on lower back
* tumor on the back
* ankylosing spondylitis
* previous lumbar surgery
* coagulopathy or bleeding tendency
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
pain intensity and interference | Data were collected using the Short Form of the Brief Pain Inventory (BPI-SF) : baseline before the intervention, and the change from pain intensity and interference at 1 month.
  Primary pain outcomes were measured by the Chinese version of the Brief Pain Inventory-Short Form (BPI-SF), which consists of 11 items to measure pain intensity and interference with functionality. Regarding pain severity, 4 items allow patients to rate their pain experience in the past 24 hours or one week at its average, worst, and least levels, as well as their pain experience now, on an 11-point Likert-type scale (0 = no pain, 10 = most severe pain).

SECONDARY OUTCOMES:
life dysfunction | Data were collected using the Roland-Morris Disability Questionnaire (RDQ) : baseline before the intervention, and the change from life dysfunction at 1 month.
  Secondary outcomes were aspects of life dysfunction as measured by the Roland Morris Disability Questionnaire (RMDQ), which measures disability in daily life due to LBP. This questionnaire consists of 24 items, each one a statement that the patient is asked to indicate whether this statement applies to him/her.

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Hua Yang, MASTER, Principal Investigator — EN CHU HOSPITAL
Locations (1):
- En Chu Kong Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang HH, Chung YC, Szeto PP, Yeh ML, Lin JG. Laser acupuncture combined with auricular acupressure improves low-back pain and quality of life in nurses: A randomized controlled trial. J Integr Med. 2023 Jan;21(1):26-33. doi: 10.1016/j.joim.2022.10.004. Epub 2022 Oct 17. PMID 36402666

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT04423445/Prot_SAP_000.pdf